CLINICAL TRIAL: NCT02321163
Title: A New Paradigm of Neuromuscular Electrical Stimulation in Attenuating Muscle Atrophy: a Randomised Controlled Trial
Brief Title: Electrical Stimulation for Attenuating Muscle Atrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Simon S. Yeung, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HMRF12131991
Record Dates: First submitted 2014-12-08; First posted 2014-12-22 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NMES new paradigm (Experimental): For the NMES new paradigm, A portable electrical stimulator will be used to produce simultaneous stimulation to both the quadriceps and calf muscles. The stimulator delivers a biphasic, asymmetrical square wave at a pulse width of 250 μs and duty cycle 5:10 sec with 2 Hz frequencies of stimulation. To disperse current intensity and enhance the comfort of the stimulation, large rectangular electrodes (80 × 100 mm) will be positioned at the best motor points of the quadriceps and calf muscles. The electrodes will be secured by tight short and sock at the respective positions. The stimulation intensity will be set to just visible muscle contractions. Stimuli will be applied twice a day for 3 h (with a 2 h rest between treatments), 5 days a week for 8 weeks.
  Interventions: Device: NMES new paradigm
- NMES conventional (Active Comparator): For NMES conventional, the experimental protocol will be the conventional electrical stimulation protocol i.e frequency: 50 Hz; intensity: maximum intensity tolerated by the subject; duration: 30 min.
  Interventions: Device: NMES conventional
- Placebo (Sham Comparator): For placebo, electrodes will be applied and all conditions will be similar to those in the NMES group, except that the amplitude will be set to 0 mA so that no muscle stimulation occurs.
  Interventions: Device: NMES no stimulation

INTERVENTIONS:
Device: NMES new paradigm — stimulation frequency: 2 Hz; intensity: low amplitude; duration: 3 hours, 2 times per day for 8 weeks
  Arms: NMES new paradigm
Device: NMES conventional — stimulation frequency: 50 Hz; intensity: maximally tolerated; duration: 30 min per day for 8 weeks
  Arms: NMES conventional
Device: NMES no stimulation — Placebo, electrode pad on, no stimulation
  Arms: Placebo

SUMMARY:
Objectives: This study aims to examine the use of low frequency (2Hz), low amplitude (intensity just produce visible muscle contraction), and long duration (2x3 hrs/day) neuromuscular electrical simulation (NMES) in attenuating the effects of muscle atrophy resulted from disuse.

Design and subjects: The study is a randomized, double-blind, controlled, and parallel group study. Subjects with stable chronic obstructive pulmonary disease (COPD) will be included. Intervention: Subjects will be randomized to 3 groups to receive different NMES program over the quadriceps and calf muscles: (i) the proposed NMES program; (ii) conventional NMES program (50Hz, 30 min/day), or sham group for a period of 8 weeks.

Outcome measures:The effectiveness of the NMES will be evaluated by the improvement in muscle cross-sectional area (CSA), muscle performance (muscle strength, muscle shortening velocity and muscle activation testing), functional performance (6 min walk) and subjects' rating of the perceived acceptability of the stimulation protocol.

Data analysis: Baseline characteristics of the intervention and sham groups will be compared using one way ANOVA. Two-way mixed repeated measures analysis of variance will be performed to examine the differences between groups over time for all the outcome variables. The significance level is set at p < 0.05.

Expected results: The investigators hypothesize that the proposed new paradigm of NMES would be more effective in improving muscle cross-sectional area (CSA), strength, endurance, and exercise tolerance.

DETAILED DESCRIPTION:
Introduction:

Skeletal muscle responds to the stimulus of mechanical load for growth and maintenance. Prolonged reductions in muscle activity and mechanical loading such as spaceflight, limb immobilization, bedrest, and/or inactivity alter the balance between protein synthesis and degradation, resulting in skeletal muscle atrophy (1-3). This is characterized by a decrease in muscle mass, myofiber cross-sectional area, contractile strength and speed, as well as slow-to-fast fiber type transformation (4,5). Many countermeasures have been reported to attenuate the loss of muscle atrophy and neuromuscular electrical stimulation (NMES) has been frequently used in conditions such as spinal cord injury, immobilization, and muscle disuse post-surgery (6,7). Indeed, a recent Cochrane review on the effectiveness of NMES for muscle weakness in adults with progressive diseases such as COPD, chronic heart failure and cancer indicated that NMES is an effective means of improving muscle weakness (8). The meta-analyses included eleven randomized controlled trial (RCT) studies involving a total of 218 participants. NMES significantly improved quadriceps strength by a Standardised Mean Difference (SMD) of 0.9 (95% confidence interval (CI) 0.33 to 1.46). This is approximately equals to 25 Newton metres (Nm) and should be regarded as clinically significant. Similarly, another recent systematic review also showed NMES is effective in preventing skeletal-muscle weakness in critically ill patients. Eight eligible studies involving 172 patients were included in the analysis. Out of the eight studies, five studies reported an increase in strength or better preservation of strength with NMES, with one study having a large effect size (1.44). Two studies found better preservation of muscle mass with NMES, with small to moderate effect sizes (0.11-0.39) while no significant benefits were found in two other studies (9).

The effectiveness of NMES is dependent upon the clinical condition and is influenced by different stimulation parameters, particularly the stimulation frequency and duration. Traditionally, NMES has been viewed as the application of a transcutaneous electrical current to the neuromuscular junction, aimed to depolarise the motor unit action potential and inducing muscle contraction (10). This electrically induced muscle contraction simulates active muscle strengthening and is based on the principle of muscle training that by appropriate loading, muscle strength will be increased. To achieve this training effect, the stimulation parameters employed normally aimed to produce tetanic contraction with a current density that the subject can maximally tolerated (8,9). However, this currently adopted stimulation protocol (ie. high frequency at or above 50Hz, amplitude at subjects' maximum tolerated limit and short duration (30 min to 1 hr) to counteract muscle atrophy has two main drawbacks. First, it has been well established that mechanical unloading is associated with detrimental changes to the structure and function of skeletal muscles, characterized by reduction in muscle mass, myofiber cross-sectional area, contractile strength and speed, as well as slow-to-fast fiber type transformation (for review, see 11). Thus, the slow twitch muscle fibers are more susceptible to unloading or disuse effect rather than fast twitch muscle fibers. The traditional high frequency stimulation protocol (50 Hz) does not match the motor unit firing pattern of a slow-twitch muscle. Moreover, the high current density would inevitably caused discomfort if not pain to the subjects during the electrical stimulation. The subjects cannot tolerate the electrical stimulation for hours. This is particularly the case if the application is to the subjects with disuse muscle atrophy or subjects with muscle weakness caused by progressive diseases. Very often, the pain tolerance of this group of subjects is generally lower than the normal healthy subjects. Thus, the currently adopted protocol might not necessary render the best possible outcome of NMES for the enhancement of muscle function. The beneficial effects of NMES to counteract muscle atrophy had not been fully utilized. A recent systematic review that examines metabolic and structural changes in lower limb skeletal muscle following neuromuscular electrical stimulation identified only 18 studies. Eight of these studies investigated enzymatic activities, seven studies on muscle fibre composition, and 14 on muscle fibre size. Among these 18 studies, only 9 are RCT studies, and the methodological quality generally was poor. The authors concluded that NMES seems to be able to produce favourable changes in oxidative enzyme activity, skeletal muscle fibre type and skeletal muscle fibre size. In view of the large heterogeneity in NMES protocols, the authors concluded that there was no definite consensus regarding the stimulation frequencies for optimal muscular changes (12), For instance, Theriault et al. (13) had conducted prolonged electrical stimulation to the knee extensor of 8 healthy adults. The electrical stimulation protocol was of 8-week duration for 8 hour per day and 6 days per week. The stimulation parameter was of low frequency (8 Hz) with intensity just being able to produce visible vibration. The results suggested significant improvement in knee extensor performance after 4 week of stimulation. However, the study is not a RCT study and there is control group in the study. On the other hand, one of the RCT studies that investigated the effects of NMES and incorporated high frequency (50Hz) but very low amplitude (without muscle contraction) as the placebo group had incidentally revealed that the placebo produced better effect than the intervention group. The NMES group vs placebo group by a SMD of -0.12 (95% CI: -0.63, 0.39) (8,14). Banerjee and his group has also shown an electrical stimulation protocol with low frequency (4 Hz) yet high amplitude (300mA), 1 hr/day for 6 week can significantly increase the quadriceps strength of healthy sedentary adults and patients with stable chronic heart failure (15, 16). Thus, the findings from basic science and these clinical studies suggested the need for further exploration of more effective NMES stimulation protocol to attenuate muscle atrophy.

Aims and Hypotheses to be Tested:

To address these, the investigators of this proposal have challenged the traditional thought that NMES should be with high frequency and high amplitude. The investigators had tested the hypothesis that low frequency and low amplitude is effective in attenuating muscle atrophy, and investigated the cellular mechanisms associated with muscle unloading. Using the hindlimb suspension animal model, the investigators have previously demonstrated that, during hindlimb suspension, application of low-frequency electrical stimulation at 20 Hz on the soleus muscles with defined timing and pulse parameters partially rescued the loss of satellite cells and improved fiber cross-sectional areas (17). The investigators have further demonstrated that using an electrical stimulation paradigm of frequency: 20 Hz; duration: 3 h, twice daily to eight-week-old male BALB/c mice that were subjected to a 14-day hindlimb unloading (HU). This stimulation paradigm can enhance satellite cell proliferative potential as well as suppress apoptotic cell death in disuse induced muscle atrophy. Morphologically, the hindlimb with electrical stimulation showed significant improvement in muscle mass, cross-sectional area, and peak tetanic force relative to the HU limb (18). Recently, the investigators further investigated the optimum stimulation protocol and demonstrated that among three low frequency protocol, 2, 10 and 20 Hz, stimulation at 2 Hz for 2 × 3 h/day achieved the best effect in attenuating the loss of muscle fiber cross-sectional area and force. This stimulation parameter led to a 1.2-fold increase in satellite cell proliferation, and was effective in rescuing cells from apoptosis (19). With all these encouraging findings from the basic science research, the investigators believe the proposed new paradigm of NMES can be tested on subjects with progressive muscle atrophy. The investigators hypothesis that NMES at 2 Hz for 2 × 3 h/day is effective in attenuating/improving lower limb postural muscle atrophy, namely quadriceps and gastrocnemius and soleus muscle complex.

Plan of Investigation:

Based on the findings in the existing literature on the current adopted NMES stimulation protocol in attenuating muscle atrophy or improving muscle performance in various populations, the investigators hypothesized that the proposed new paradigm of NMES would be more effective in improving muscle cross-sectional area (CSA), strength, endurance, exercise tolerance, and is more acceptable by subjects who needed NMES to attenuating the muscle atrophy with various medical conditions, in particular chronic obstructive pulmonary disease (COPD) patients.

ELIGIBILITY:
Inclusion Criteria:

* stable COPD patients who had been discharged from the medical unit, and had been admitted less than 2 times in the preceding year;
* patients drawn from either pulmonary rehabilitation program in Day Care Centre; or self help group; or home bound;
* COPD subjects with Forced Expiratory Volume at 1 sec (FEV1) to Forced Vital Capacity (FVC) ratio: ≤ 70%, oxygen uptake maximum (VO2 max) ≤ 8 MET and BMI ≤ 21kg/m2

Exclusion Criteria:

* subjects with known muscle wasting diseases such as motor neuron disease, cachexia, e.g. cancer cachexia;
* subjects with muscle dysfunction as a result of neurological conditions such as stroke, Parkinsonism
* subjects that can not comply with the study procedures (e.g. dementia)

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-12 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Muscle cross sectional area (quadriceps and calf muscles) | 8 weeks
  Ultrasonography of the quadriceps and calf muscle cross sectional area measured at baseline, week 4 and week 8 of the study.

SECONDARY OUTCOMES:
Isometric knee extensor and plantarflexor muscle torque | 8 weeks
  The maximum isometric peak torque of knee extensor and plantarflexor measured at baseline, week 4 and week 8 of the study.
Muscle activation (Twitch interpolation technique will be used to assess the voluntary muscle activation) | 8 weeks
  Twitch interpolation technique will be used to assess the voluntary muscle activation of the quadriceps and calf muscles at baseline, week 4 and week 8 of the study.
Functional ability (improvement of the muscle strength will furthered be tested on the 6-min walk test) | 8 weeks
  The improvement of the muscle strength will furthered be tested on the 6-min walk test. The walking distance will be measured at baseline, week 4 and week 8 of the study.
Acceptability of the stimulation protocol (10 point scale) | 8 weeks
  A 10 point scale will be used for the subjects to rate the extent of discomfort associated with the stimulation protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Simon S Yeung, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Department of Rehabilitation Sciences, The Hong Kong Polytechnic University, Hung Hom, Hong Kong

REFERENCES:
- [Background] Paddon-Jones D, Sheffield-Moore M, Cree MG, Hewlings SJ, Aarsland A, Wolfe RR, Ferrando AA. Atrophy and impaired muscle protein synthesis during prolonged inactivity and stress. J Clin Endocrinol Metab. 2006 Dec;91(12):4836-41. doi: 10.1210/jc.2006-0651. Epub 2006 Sep 19. PMID 16984982
- [Background] Greenhaff PL. The molecular physiology of human limb immobilization and rehabilitation. Exerc Sport Sci Rev. 2006 Oct;34(4):159-63. doi: 10.1249/01.jes.0000240017.99877.8a. PMID 17031253
- [Background] Fitts RH, Riley DR, Widrick JJ. Functional and structural adaptations of skeletal muscle to microgravity. J Exp Biol. 2001 Sep;204(Pt 18):3201-8. doi: 10.1242/jeb.204.18.3201. PMID 11581335
- [Background] Fitts RH, Riley DR, Widrick JJ. Physiology of a microgravity environment invited review: microgravity and skeletal muscle. J Appl Physiol (1985). 2000 Aug;89(2):823-39. doi: 10.1152/jappl.2000.89.2.823. PMID 10926670
- [Background] Adams GR, Caiozzo VJ, Baldwin KM. Skeletal muscle unweighting: spaceflight and ground-based models. J Appl Physiol (1985). 2003 Dec;95(6):2185-201. doi: 10.1152/japplphysiol.00346.2003. PMID 14600160
- [Background] Sheffler LR, Chae J. Neuromuscular electrical stimulation in neurorehabilitation. Muscle Nerve. 2007 May;35(5):562-90. doi: 10.1002/mus.20758. PMID 17299744
- [Background] Bax L, Staes F, Verhagen A. Does neuromuscular electrical stimulation strengthen the quadriceps femoris? A systematic review of randomised controlled trials. Sports Med. 2005;35(3):191-212. doi: 10.2165/00007256-200535030-00002. PMID 15730336
- [Background] Maddocks M, Gao W, Higginson IJ, Wilcock A. Neuromuscular electrical stimulation for muscle weakness in adults with advanced disease. Cochrane Database Syst Rev. 2013 Jan 31;(1):CD009419. doi: 10.1002/14651858.CD009419.pub2. PMID 23440837
- [Background] Maffiuletti NA, Roig M, Karatzanos E, Nanas S. Neuromuscular electrical stimulation for preventing skeletal-muscle weakness and wasting in critically ill patients: a systematic review. BMC Med. 2013 May 23;11:137. doi: 10.1186/1741-7015-11-137. PMID 23701811
- [Background] Petterson S, Snyder-Mackler L. The use of neuromuscular electrical stimulation to improve activation deficits in a patient with chronic quadriceps strength impairments following total knee arthroplasty. J Orthop Sports Phys Ther. 2006 Sep;36(9):678-85. doi: 10.2519/jospt.2006.2305. PMID 17017273
- [Background] Sillen MJ, Franssen FM, Gosker HR, Wouters EF, Spruit MA. Metabolic and structural changes in lower-limb skeletal muscle following neuromuscular electrical stimulation: a systematic review. PLoS One. 2013 Sep 3;8(9):e69391. doi: 10.1371/journal.pone.0069391. eCollection 2013. PMID 24019860
- [Background] Theriault R, Theriault G, Simoneau JA. Human skeletal muscle adaptation in response to chronic low-frequency electrical stimulation. J Appl Physiol (1985). 1994 Oct;77(4):1885-9. doi: 10.1152/jappl.1994.77.4.1885. PMID 7836213
- [Background] Napolis LM, Dal Corso S, Neder JA, Malaguti C, Gimenes AC, Nery LE. Neuromuscular electrical stimulation improves exercise tolerance in chronic obstructive pulmonary disease patients with better preserved fat-free mass. Clinics (Sao Paulo). 2011;66(3):401-6. doi: 10.1590/s1807-59322011000300006. PMID 21552662
- [Background] Banerjee P, Caulfield B, Crowe L, Clark AL. Prolonged electrical muscle stimulation exercise improves strength, peak VO2, and exercise capacity in patients with stable chronic heart failure. J Card Fail. 2009 May;15(4):319-26. doi: 10.1016/j.cardfail.2008.11.005. Epub 2009 Jan 29. PMID 19398080
- [Background] Banerjee P, Caulfield B, Crowe L, Clark A. Prolonged electrical muscle stimulation exercise improves strength and aerobic capacity in healthy sedentary adults. J Appl Physiol (1985). 2005 Dec;99(6):2307-11. doi: 10.1152/japplphysiol.00891.2004. Epub 2005 Aug 4. PMID 16081619
- [Result] Zhang BT, Yeung SS, Liu Y, Wang HH, Wan YM, Ling SK, Zhang HY, Li YH, Yeung EW. The effects of low frequency electrical stimulation on satellite cell activity in rat skeletal muscle during hindlimb suspension. BMC Cell Biol. 2010 Nov 18;11:87. doi: 10.1186/1471-2121-11-87. PMID 21087483
- [Result] Guo BS, Cheung KK, Yeung SS, Zhang BT, Yeung EW. Electrical stimulation influences satellite cell proliferation and apoptosis in unloading-induced muscle atrophy in mice. PLoS One. 2012;7(1):e30348. doi: 10.1371/journal.pone.0030348. Epub 2012 Jan 12. PMID 22253929